CLINICAL TRIAL: NCT06897033
Title: Effect of Artificial Intelligence-Generated WhatsApp Reminders Compared to No Reminders on Oral Health Among Young Adults: A Randomized Controlled Trial
Brief Title: AI-Generated WhatsApp Reminders vs. No Reminders: Impact on Oral Health in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Kamel, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPER 1-3-2
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: White Spot Lesions; Dental Plaque; Oral Hygiene, Oral Health
Keywords: Oral hygiene; Reminders
MeSH Terms: conditions — Dental Plaque | interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To maintain blinding in my study, I will implement the following steps:
  Supervisor-Managed Allocation: My supervisor will independently assign participants to either the intervention or control group. Each participant will receive a unique code corresponding to their group assignment, ensuring I remain unaware of their allocation.
  Automated Messaging System: I will set up an automated system to send WhatsApp reminders based on the codes assigned. This system will operate without revealing to me which participants receive the messages, preserving the blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Education followed by Whatsapp AI-Generated Reminders Group (Experimental): This arm will receive oral health education followed by Whatsapp AI-generated text messages as reminders design to motivate, uplift self efficacy and remind individuals to practice good oral hygiene measures over the course of 3 months.
  Interventions: Behavioral: Health education followed by AI-generated Whatsapp reminders; Behavioral: Oral Health Education
- Health Education Only (Active Comparator): This group will receive personal health education session only.
  Interventions: Behavioral: Oral Health Education

INTERVENTIONS:
Behavioral: Health education followed by AI-generated Whatsapp reminders — Participants will receive dental health education in a one to one personal session followed by Text messages generated by AI large language model (ChatGPT free version) about oral hygiene practices for three month in a tapering frequency. These messages will be designed based on Fogg's Behavior Model, focusing on enhancing motivation, ability, and providing clear triggers for action.
  Arms: Health Education followed by Whatsapp AI-Generated Reminders Group
Behavioral: Oral Health Education — Oral health education in a one to one session explaining the importance of oral hygiene measures and demonstrating teeth brushing techniques and healthy dietary guidelines and recommendations.

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of artificial intelligence-generated WhatsApp reminders on improving oral hygiene practices among individuals aged 20-40 years visiting the periodontal clinic at El-Qasr El-Ainy Dental Hospital. Participants will be randomly assigned to either receive health education followed by AI-generated WhatsApp reminders over a 3-month period or to a control group receiving health education only. The primary outcome is the presence of white spot lesions, assessed using the modified Gorelick White Spot Lesion (WSL) index. Secondary outcomes include the presence of dental plaque, measured by the Plaque Index (PI). This study seeks to determine whether AI-generated reminders can enhance oral hygiene adherence compared to standard health education alone.

ELIGIBILITY:
Inclusion Criteria:

* Received a non-surgical periodontal treatment and oral hygiene instructions.
* Own a smartphone with WhatsApp installed.
* Willing and able to provide informed consent to participate in the study.

Exclusion Criteria:

* Individuals with pre-existing oral health conditions requiring specialized care.
* Patients who received surgical periodontal interventions.
* Participation in another oral health or diet-related study.
* Individuals who do not use WhatsApp or are unwilling to receive messages through the platform.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
White Spot Lesion in the oral cavity | 3 Months
  Presence of white spot lesions which will be measured by the modified Gorelick WSL index (Gorelick et al., 1982) which uses categorical scoring system from 0-3.

SECONDARY OUTCOMES:
Presence of Plaque | 3 Months
  Presence of dental plaque which will be measured using the Plaque Index (PI) (Silness & Löe, 1964) measured as percentage (%) of tooth surfaces with plaque.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Abou El Fadl RK, Abdel Fattah MA, Helmi MA, Wassel MO, Badran AS, Elgendi HAA, Allam MEE, Mokhtar AG, Saad Eldin M, Ibrahim EAY, Elgarba BM, Mehlis M. Periodontal diseases and potential risk factors in Egyptian adult population-Results from a national cross-sectional study. PLoS One. 2021 Nov 3;16(11):e0258958. doi: 10.1371/journal.pone.0258958. eCollection 2021. PMID 34731192
- [Background] Albandar JM, Rams TE. Global epidemiology of periodontal diseases: an overview. Periodontol 2000. 2002;29:7-10. doi: 10.1034/j.1600-0757.2002.290101.x. No abstract available. PMID 12102700
- [Background] Brigden A, Anderson E, Linney C, Morris R, Parslow R, Serafimova T, Smith L, Briggs E, Loades M, Crawley E. Digital Behavior Change Interventions for Younger Children With Chronic Health Conditions: Systematic Review. J Med Internet Res. 2020 Jul 31;22(7):e16924. doi: 10.2196/16924. PMID 32735227
- [Background] Eppright M, Shroff B, Best AM, Barcoma E, Lindauer SJ. Influence of active reminders on oral hygiene compliance in orthodontic patients. Angle Orthod. 2014 Mar;84(2):208-13. doi: 10.2319/062813-481.1. Epub 2013 Sep 12. PMID 24028316
- [Background] Fogg BJ. A behavior model for persuasive design. Proceedings of the 4th International Conference on Persuasive Technology. New York: ACM; 2009. p. 40.
- [Background] Gentili A, Failla G, Melnyk A, Puleo V, Tanna GLD, Ricciardi W, Cascini F. The cost-effectiveness of digital health interventions: A systematic review of the literature. Front Public Health. 2022 Aug 11;10:787135. doi: 10.3389/fpubh.2022.787135. eCollection 2022. PMID 36033812
- [Background] Kumar GS, Kashyap A, Raghav S, Bhardwaj R, Singh A, Guram G. Role of Text Message Reminder on Oral Hygiene Maintenance of Orthodontic Patients. J Contemp Dent Pract. 2018 Jan 1;19(1):98-101. doi: 10.5005/jp-journals-10024-2219. PMID 29358543
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Mekhemar M, Ebeid K, Attia S, Dorfer C, Conrad J. Oral Health Attitudes among Preclinical and Clinical Dental Students: A Pilot Study and Self-Assessment in an Egyptian State-Funded University. Int J Environ Res Public Health. 2020 Dec 30;18(1):234. doi: 10.3390/ijerph18010234. PMID 33396877
- [Background] Orth M, Averina M, Chatzipanagiotou S, Faure G, Haushofer A, Kusec V, Machado A, Misbah SA, Oosterhuis W, Pulkki K, Twomey PJ, Wieland E. Opinion: redefining the role of the physician in laboratory medicine in the context of emerging technologies, personalised medicine and patient autonomy ('4P medicine'). J Clin Pathol. 2019 Mar;72(3):191-197. doi: 10.1136/jclinpath-2017-204734. Epub 2017 Dec 22. PMID 29273576
- [Background] Pubalan S, Zi Hong O, Yongxian T, Mabel L. Assessing effectiveness of WhatsApp messaging program in oral hygiene care for orthodontic patients: A randomised controlled trial. J Orthod. 2024 Dec;51(4):407-414. doi: 10.1177/14653125241230561. Epub 2024 Feb 17. PMID 38366912
- [Background] Ross MC, Campbell PM, Tadlock LP, Taylor RW, Buschang PH. Effect of automated messaging on oral hygiene in adolescent orthodontic patients: A randomized controlled trial. Angle Orthod. 2019 Mar;89(2):262-267. doi: 10.2319/040618-260.1. Epub 2018 Dec 5. PMID 30516416
- [Background] Samvel Mkhitaryan, Philippe J. Giabbanelli, Nanne K. de Vries, Rik Crutzen. Dealing with complexity: How to use a hybrid approach to incorporate complexity in health behavior interventions. Intelligence-Based Medicine. 2020; 3-4: 1-13.
- [Background] Saxena K, Gunjal S. Influence of WhatsApp and electronic mail reminders on oral hygiene compliance of orthodontic patients using planimetry : A randomized clinical trial. J Orofac Orthop. 2022 Jul;83(4):269-276. doi: 10.1007/s00056-021-00301-6. Epub 2021 May 4. PMID 33944974
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] 17. Splieth CH. Prevention of periodontal disease in children and adolescents. Int J Paediatr Dent. 2005 Jan;15(1):7-13.
- [Background] Senocak I, Camci H. Effect of various active reminders via mobile phone on cooperation of orthodontic teenage patients regarding oral hygiene and Class II elastics use : A three-month follow-up prospective cohort study. J Orofac Orthop. 2025 Aug;86(Suppl 1):39-47. doi: 10.1007/s00056-024-00549-8. Epub 2024 Sep 14. PMID 39276182